CLINICAL TRIAL: NCT05573698
Title: A Phase 1b, Randomized, Double-blind, Placebo-controlled, Multiple Ascending Dose and Multi-Dose Study of DT-216 in Adult Patients With Friedreich Ataxia
Brief Title: Study to Evaluate Multiple Ascending Dose and Multi-Dose of DT-216 in Adult Patients With Friedreich Ataxia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Design Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DTX-216-102
Record Dates: First submitted 2022-10-06; First posted 2022-10-10 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Friedreich Ataxia
MeSH Terms: conditions — Friedreich Ataxia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Multiple Dose: DT-216 (Experimental): Participants will be administered multiple doses of DT-216
  Interventions: Drug: DT-216
- Multiple Dose: DT-216 matching placebo (Placebo Comparator): Participants will be administered multiple doses of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DT-216 — DT-216 will be administered by intravenous (IV) injection
  Arms: Multiple Dose: DT-216
Drug: Placebo — Matching Placebo will be administered by intravenous (IV) injection
  Arms: Multiple Dose: DT-216 matching placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetic, and pharmacodynamic effects of multiple doses of intravenous DT-216 in adult patients with Friedrich Ataxia.

ELIGIBILITY:
Inclusion Criteria:

* Genetically confirmed diagnosis of Friedreich Ataxia with homozygous GAA repeat expansions.
* Able and willing to sign informed consent form prior to study enrollment.
* Stage 5.5 or less on the Functional Staging for Ataxia (FSA) at screening.

Exclusion Criteria:

* Has any concomitant medical condition that in the opinion of the investigator, puts the participant at risk or precludes participant from completing the study.
* Has clinically significant abnormal laboratory results.
* Has significant cardiac disease.
* Received an investigational drug within 3 months of screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-09-27 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2023-08-25 (Actual)

PRIMARY OUTCOMES:
Safety Measure | Up to approximately 60 days
  Frequency of treatment emergent adverse events (TEAEs)

SECONDARY OUTCOMES:
Pharmacokinetic parameters | Up to approximately 60 days
  Maximum Plasma Concentration (Cmax) of DT-216
Pharmacokinetic parameters | Up to approximately 60 days
  Time to Maximum Plasma Concentration (Tmax) of DT-216
Pharmacokinetic parameters | Up to approximately 60 days
  Area Under the Concentration-time Curve (AUC) of DT-216

OTHER OUTCOMES:
Pharmacodynamic parameters | Up to approximately 60 days
  Frataxin expression

CONTACTS AND LOCATIONS:
Locations (1):
- Clinilabs, Eatontown, New Jersey, United States